CLINICAL TRIAL: NCT05659927
Title: Safety, Tolerability, and Pharmacokinetics of MG-ZG122 in a Single Subcutaneous Injection in Chinese Healthy Adult Subjects: a Single-center, Randomized, Double-blind, Placebo-controlled, Dose-increasing Phase I Clinical Trial
Brief Title: Single Dose Clinical Trial of MG-ZG122 in Chinese Healthy Adult Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Mabgeek Biotech.Co.Ltd (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MG-ZG122-01
Record Dates: First submitted 2022-11-24; First posted 2022-12-21 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Intervention Model Description: Subcutaneous injections were 52.5 mg, 105 mg, 210 mg and 420 mg, respectively. Four patients were included in the 52.5 mg dose group (2 in the drug group and 2 in the placebo group). There were 10 cases in the other 3 dose groups (8 cases in the drug group and 2 cases in the placebo group). In accordance with the principle of dose increment, from low dose to high dose.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MG-ZG122 first dose group (Experimental): 4 cases in the 52.5 mg dose group (2 cases of placebo, 2 cases of experimental drug)
  Interventions: Drug: MG-ZG122 Humanized Monoclonal Antibody Injection; Drug: Placebo
- MG-ZG122 second dose group (Experimental): 10 cases in the 105 mg dose group (2 cases of placebo, 8 cases of experimental drug)
  Interventions: Drug: MG-ZG122 Humanized Monoclonal Antibody Injection; Drug: Placebo
- MG-ZG122 third dose group (Experimental): 10 cases in the 210 mg dose group (2 cases of placebo, 8 cases of experimental drug)
  Interventions: Drug: MG-ZG122 Humanized Monoclonal Antibody Injection; Drug: Placebo
- MG-ZG122 forth dose group (Experimental): 10 cases in the 420 mg dose group (2 cases of placebo, 8 cases of experimental drug)
  Interventions: Drug: MG-ZG122 Humanized Monoclonal Antibody Injection; Drug: Placebo

INTERVENTIONS:
Drug: MG-ZG122 Humanized Monoclonal Antibody Injection — Single subcutaneous injection. Subjects with a dose of less than or equal to 2 ml were given one injection, and subjects with a dose of more than 2 ml were given two injections. A group 0.5 ml, B group 1 ml, C group 2 ml, D group 4 ml.
  Other Names: MG-ZG122
Drug: Placebo — Single subcutaneous injection. Subjects with a dose of less than or equal to 2 ml were given one injection, and subjects with a dose of more than 2 ml were given two injections. A group 0.5 ml, B group 1 ml, C group 2 ml, D group 4 ml.

SUMMARY:
To determine the safety and tolerability of MG-ZG122 in Chinese healthy adult subjects

DETAILED DESCRIPTION:
Main purpose: To determine the safety and tolerability of MG-ZG122 humanized monoclonal antibody injection (MG-ZG122 for short) in Chinese healthy adult subjects.

Secondary objective: To study the pharmacokinetic (PK) characteristics of MG-ZG122 in healthy Chinese adult volunteers, and to provide a basis for the design of clinical trial protocols for subsequent clinical trials; To evaluate the immunogenicity of MG-ZG122 in Chinese healthy adult volunteers; Preliminary exploration of the efficacy of MG-ZG122 in Chinese healthy adult subjects Impact of Biomarkers in Physiology (PD).

ELIGIBILITY:
Inclusion Criteria:

- 1. The subjects signed the ICF before the study and fully understood the research content, process and possible adverse reactions; voluntarily participated in the study and were able to complete the study according to the program requirements.

2. Chinese healthy adult subjects aged 18-65 years (including the boundary value) , both male and female; 3. Male volunteers weighing ≥50 kg; women weighing ≥40 kg; body mass index (BMI) within the range of 19.0-26.0 kg/m2 (including boundary values; BMI=weight kg/height 2 m2);

Exclusion Criteria:

1. Patients with acute or subacute infection (such as fever, cough, urgency, dysuria, abdominal pain, diarrhea and skin infection wounds, etc.) within 2 weeks before screening, or acute or chronic infection within 4 weeks before screening history, and receiving systemic anti-infective treatment;
2. Those who have a history of tuberculosis infection in the past;
3. The results of physical examination, vital sign measurement, laboratory examination, electrocardiogram, chest X-ray, etc. are abnormal and have clinical significance;
4. Those who are known to be allergic to monoclonal antibody drugs or excipients of MG-ZG122 injection, or food allergies judged by the investigator to be unsuitable to participate in the researcher;
5. Those who have been vaccinated within 1 month before screening or plan to be vaccinated during the study;
6. Those who have used any prescription drugs within 2 weeks before administration, those who have used non-prescription drugs or traditional Chinese medicines within 1 week before administration, or those who are expected to use prescription drugs, non-prescription drugs and traditional Chinese medicines during the study period;
7. Those who have received any research non-biological agents within 5 half-lives (if known) or within 3 months (whichever is longer) before administration, or have participated in other clinical trials or plan to participate in other clinical trials during the study period. clinical trial subjects;
8. Those who have special requirements for diet or cannot accept a unified diet;
9. Women who are lactating and pregnant, or female volunteers of childbearing age have a positive serum pregnancy test;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2024-01-26 (Actual); Study Completion 2024-03-23 (Estimated)

PRIMARY OUTCOMES:
Tolerability and Safety Analysis | up to 127 days
  Evaluate for dose escalation for study termination criteria or achievement of MTD

SECONDARY OUTCOMES:
Pharmacokinetic Analysis of Cmax | 127 days
  Evaluate the pharmacokinetic parameters Cmax of MG-ZG122
Pharmacokinetic Analysis of Tmax | 127 days
  Evaluate the pharmacokinetic parameters Tmax of MG-ZG122
Pharmacokinetic Analysis of AUC0-t | 127 days
  Evaluate the pharmacokinetic parameters AUC0-t of MG-ZG122
Pharmacokinetic Analysis of t1/2 | 127 days
  Evaluate the pharmacokinetic parameters t1/2 of MG-ZG122
Pharmacokinetic Analysis of AUC0-∞ | 127 days
  Evaluate the pharmacokinetic parameters AUC0-∞ of MG-ZG122
Pharmacodynamic Biomarker Analysis of serum interleukin-5 | 127 days
  The effect of MG-ZG122 was evaluated by the changes of serum interleukin-5 before and after administration at each follow-up time point
Pharmacodynamic Biomarker Analysis of immunoglobulin E | 127 days
  The effect of MG-ZG122 was evaluated by the changes of immunoglobulin E (Immunoglobulin E, IgE) before and after administration at each follow-up time point
Pharmacodynamic Biomarker Analysis of the number of eosinophils in peripheral blood | 127 days
  The effect of MG-ZG122 was evaluated by the changes of the number of eosinophils in peripheral blood before and after administration at each follow-up time point
Immunogenicity ADA | 127 days
  Antidrug Antibody (ADA) Incidence (if applicable) and Their Impact on PK, Safety, and Efficacy
Neutralizing Antibody (Nab) | 127 days
  Neutralizing Antibody (Nab) IncidenceIncidence (if applicable) and Their Impact on PK, Safety, and Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zhao, Principal Investigator — The Second Hospital of Anhui Medical University; Wei Hu, Principal Investigator — The Second Hospital of Anhui Medical University
Locations (1):
- The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No
We may work with other companies to develop follow-up clinical programs in China or global clinical programs

REFERENCES:
- [Derived] Zhang X, Zhu L, Zhang Q, Zheng L, Guo J, Zou Q, Yan R, Qin D, Zhang C, Hu W. Safety, tolerability, pharmacokinetics, immunogenicity, and pharmacodynamics of MG-ZG122, a long-acting humanized anti-thymic stromal lymphopoietin mAb, in healthy Chinese: a randomized, double-blind, placebo-controlled, dose-escalation, phase I study. Expert Opin Investig Drugs. 2025 Nov;34(11):943-951. doi: 10.1080/13543784.2025.2581666. Epub 2025 Oct 30. PMID 41144273